CLINICAL TRIAL: NCT03236103
Title: AKI Prevention and Early Intervention in VAD Patients Admitted for Acute Medical Events.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Qi Qian, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-002670
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury
Keywords: Ventricular assist device
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Open label single group interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with VAD in place (Other): Adult patients with VAD in place who are admitted to the hospital for acute medical illness. The investigators will provide clinical recommendations to the subject's primary care provider.
  Interventions: Other: Clinical Recommendations

INTERVENTIONS:
Other: Clinical Recommendations — The clinical recommendations will regard the following:
  1. Avoidance of potentially nephrotoxic medications (e.g. NSAIDs, intravascular contrast, nephrotoxic antimicrobials)
  2. Optimizing volume status (avoidance of volume overload or depletion)
  3. Optimizing electrolytes and acid-base status
  4. Optimizing hemodynamics (Mean arterial BP>65mmHg)
  5. Assessment of kidney function with serum creatinine and/or cystatin C
  None of the suggestions will be experimental. All suggestions will be based on standard nephrology practice.

SUMMARY:
The investigators are doing this research to investigate whether multifaceted preventive measures for newly hospitalized ventricular assist device (VAD) patients will reduce the Acute Kidney Injury (AKI) occurrence rate, progression and associated complications

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether preventive measures for newly hospitalized ventricular assist device (VAD) patients will reduce the Acute Kidney Injury (AKI) occurrence rate, progression and associated complications

Participants will be in the study for the first 7 days of hospitalization. The study investigators will access the electronic medical record daily from admission day 1 through admission day 7 in order to provide clinical recommendations in an effort to minimize AKI risk as per routine practice.

If the patient is discharged prior to day 7 the study, intervention will be terminated on day of discharge.

The investigators will review the participant's medical record up to one year after surgery.

This study will not include any experimental laboratory tests or experimental medication.

The clinical recommendations will regard the following:

1. Avoidance of potentially nephrotoxic medications (e.g. NSAIDs, intravascular contrast, nephrotoxic antimicrobials)
2. Optimizing volume status (avoidance of volume overload or depletion)
3. Optimizing electrolytes and acid-base status
4. Optimizing hemodynamics (Mean arterial BP>65mmHg)
5. Assessment of kidney function with serum creatinine and/or cystatin C None of the suggestions will be experimental. All suggestions will be based on standard nephrology practice.

The investigators plan to compare the results of the current study with those in in the years of 2012-2017 (1/7/2012- 1/7/2017) via retrospective chart review

ELIGIBILITY:
Inclusion criteria:

Adult patients with VAD in place who are admitted to the hospital for acute medical illness during the study period. For those with multiple admissions during the study period only the first admission will be studied.

Patients who are able to give consent. In case of patients that are mentally impaired we will obtain consent from power of attorney and when patients regain intact mental capacity we will reobtain consent from the patient.

Exclusion criteria:

Patients on dialysis (hemodialysis or peritoneal dialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Rate of AKI in hospitalized VAD patients based on AKIN criteria | The first 7 days of hospitalization
  The AKIN staging system has 3 stages: 1) serum creatinine increase ≥ 26.5 umol/L or increase to 1.5-2.0 fold from baseline, OR urine output <0.5 ml/kg/h for 6 h; 2) serum creatinine increase > 2.0-3.0 fold from baseline OR urine output <0.5 ml/kg/h for 12 h; 3) serum creatinine increase >3.0 fold from baseline OR serum creatinine ≥354 umol/l with an acute increase of at least 44 umol/l or need for Renal Replacement Therapy (RRT) OR urine output <0.3 ml/kg/h for 24 h OR anuria for 12 OR need for RRT
Severity of AKI based on AKIN stages (I, II, III) 1 | The first 7 days of the hospitalization
  The AKIN staging system has 3 stages: 1) serum creatinine increase ≥ 26.5 umol/L or increase to 1.5-2.0 fold from baseline, OR urine output <0.5 ml/kg/h for 6 h; 2) serum creatinine increase > 2.0-3.0 fold from baseline OR urine output <0.5 ml/kg/h for 12 h; 3) serum creatinine increase >3.0 fold from baseline OR serum creatinine ≥354 umol/l with an acute increase of at least 44 umol/l or need for Renal Replacement Therapy (RRT) OR urine output <0.3 ml/kg/h for 24 h OR anuria for 12 OR need for RRT

SECONDARY OUTCOMES:
Length of hospital stay | One year after hospitalization
  The length of hospital stay will be determined from the electronic medical record.
In hospital, 60 day and one-year mortality | One year after enrollment
  The number of subjects who died during hospitalization, 60 days after hospitalization and one year after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Qi Qian, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials